CLINICAL TRIAL: NCT03594643
Title: Electronic Cigarette and Perianesthesia : a Prospective Multicentric Survey
Brief Title: Electronic Cigarette and Surgery (ECigarSurg)
Acronym: ECigarSurg
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, MD,PhD, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: 2017-Ecig-Nimes
Record Dates: First submitted 2017-12-28; First posted 2018-07-20 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Smoke Inhalation
Keywords: electronic; surgery; outcome; anesthesia; cigarette
MeSH Terms: conditions — Smoke Inhalation Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- electronic cigarette: patient using electronic device, electronic cigarette
- control: patient not smoking nor using electronic cigarette

SUMMARY:
Since decades, literature has shown that smoking has negative effect on postoperative outcome. Recent systematic review and meta-analysis on clinical impact of smoking and smoking cessation showed that postoperative healing complications occur more often in smokers compared with nonsmokers.

The use of electronic cigarette (e-cigarette) is spreading through the world. Despite this fact, the health risk assessment studies on e-cigarette are limited and scientific evidences are inconsistent.

This prospective multicenter study aimed at assessing the use of e-cigarette whether patient undergoing elective surgery. The main objective of this study was to evaluate the prevalence of e-cigarette consumer in perioperative period. Secondary objectives were to analyze when patients consume e-cigarette in regard of surgery, how many dose they consume and if they also consume nicotine cigarette.

DETAILED DESCRIPTION:
this study used a standardized questionnaire that was filled in preoperative period

ELIGIBILITY:
Inclusion Criteria:

* protocol approval
* patients scheduled for elective surgery

Exclusion Criteria:

* < 18 ans
* refusal
* not speaking
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - This study include patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
electronic cigarette | 1 day
  incidence of electronic cigarette that are used by patients

CONTACTS AND LOCATIONS:
Overall Officials: jean.yves. Lefrant, MD,PhD, Study Chair — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Cuvillon, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No